CLINICAL TRIAL: NCT04978441
Title: The Influence of Personality Characteristics and Emotions on Blood Glucose Levels Among Type 1 Diabetes Mellitus Patients
Status: Completed | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Rambam Health Care Campus (Other); Tel Aviv University (Other)
Responsible Party: Sponsor
Other Study IDs: 0436-19-TLV
Record Dates: First submitted 2021-03-02; First posted 2021-07-27 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-03

CONDITIONS: Diabetes Mellitus, Type 1; Emotions; Personality; Sleep
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Type 1 diabetes mellitus (T1DM): 1. Males or females above 18 years old
  2. Patients with a prior medical history diagnosis of T1DM
  3. Patients who are using a continuous glucose monitor (CGM or FGM)

SUMMARY:
The research goal is to find a correlation between patient personality characteristics, patients' mood and glycemic control. Eventually, using this information may allow treating physicians the ability to better balance glucose blood levels in patients with T1DM, by recognizing influencing psychological parameters. The conclusion from this research will add to other physiological parameters that are being studied today, and in the future will be integrated into an artificial pancreas.

The investigators believe that there is a correlation that hasn't been studied in the past between personality characteristics, daily emotions and the ability to balance glucose blood levels in patients with T1DM.

DETAILED DESCRIPTION:
Background:

Type 1 diabetes mellitus (T1DM), is an autoimmune disease in which cells from the immune system attack the beta cells, that produce insulin, in the pancreas. As a result of the subsequent complete insulinopenia, glycemic levels rise, and the patient completely relies on exogenous administration of sub-cutaneous insulin injections. The patients must adjust the amount of insulin along the day in accordance with measured glucose blood levels and their activities (eating, physical activity, etc.) Recently patients diagnosed with T1DM, are eligible for a continuous glucose monitor with FLASH technology (Freestyle Libre glucose monitor), within the Israeli health medical basket services. As a result, nowadays treating physicians can better monitor glucose blood levels during the day. The Freestyle Libre constantly measures subcutaneous glucose levels, translating them using a specifically designed algorithm to projected blood glucose levels. This allows for improved glycemic control and more accurate insulin dosing decisions for the patient with a tool to assess disease severity and control for the treating physician.

Using advanced algorithms, there is an enormous research effort in order to create an artificial pancreas- a glucose blood level monitor that informs an insulin pump regarding the amount of insulin that should be injected throughout the day. This will replace the patients ongoing burden of managing their glycemic levels and reduce patient dosing errors. In order to improve the already existing algorithms, inserting additional parameters into the equation may improve the predictive value of the algorithms, and thus improve the ability to balance glycemic levels in different situations. So far, most of the research in this area was performed using physiological parameters (heart rate, physical activity, nutrition, etc.).

In the suggested study the researchers wish to examine the influence of character and emotions on glycemic levels during the day. Finding a correlation between the mental and mood status and glycemia may allow for the creation of a more accurate algorithm, to better predict and balance glycemic levels in patients with T1DM.

Research hypothesis:

The investigators' hypothesis is that there is a significant correlation between baseline personality characteristics, changing emotions throughout the day, and glycemic levels in patients with T1DM.

Research goal:

The research goal is to find a correlation between patient personality characteristics, patients' mood, and glycemic control. Eventually, using this information may allow treating physicians the ability to better balance glucose blood levels in patients with T1DM, by recognizing influencing psychological parameters. The conclusion from this research will add to other physiological parameters that are being studied today, and in the future will be integrated into an artificial pancreas.

The investigators believe that there is a correlation that hasn't been studied in the past between personality characteristics, daily emotions, and the ability to balance glucose blood levels in patients with T1DM.

Methods:

During the first visit, participants will receive an explanation of nature, duration, and side effects required during the research period.

After signing the informed consent, the following information will be collected:

* Demographic and socioeconomic background
* Personality characteristics questionnaire
* Medical history including the most recent blood tests During that visit, the participant will download a designated application for his mobile device and will receive instructions on using it.

The duration of the follow-up period will be a week. During that period the patient will not change their current treatment or lifestyle. The patient will report their emotions, treatment, physical activity, behavior, and nutrition using a specifically designed smartphone application.

At the end of the data collection week, and following their next visit to the clinic, glycemic information will be downloaded from the patients' CGM/FGM device.

The mobile application: the designated application, will be built specifically for the study. The application is a questionnaire that is always available to the patient, in an accessible manner.

Through the application, the patient will be able to fill out the questionnaire at any time, asking participants for details about their mood and emotions at the time. In addition, the app will collect data, if the participant will confirm it, which is collected by the smart device (steps, pulse, etc.) The data will be stored on a computer that is locked with a password, there will be complete separation between the patient's identifying data and the research related data. Data analysis will include correlation studies between the different parameters collected- specifically looking for emotional patterns/ events that affect glycemia.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females above 18 years old
2. Patients with a prior medical history diagnosis of T1DM
3. Patients who are using a continuous glucose monitor (CGM or FGM)

Exclusion Criteria:

1. Patients without a diagnosis of type 1 DM
2. patients who are not using a continuous glucose monitor (CGM or FGM)
3. patients who did not sign an informed consent
4. lack of judgment and underage populations
5. Patients without a mobile smart device (smart phone)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a type 1 Diabetes Mellitus diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
correlation between baseline personality characteristics, changing emotions throughout the day, and glycemic levels in patients with T1DM | through study completion, an average of 1 year
  correlation between patient personality characteristics, patients' mood and glycemic control. Eventually, using this information may allow us the ability to better balance glucose blood levels in patients with T1DM, by recognizing influencing psychological parameters

CONTACTS AND LOCATIONS:
Overall Officials: Gon Shoham, MD, Study Director — Tel Aviv University
Locations (1):
- The Institute of Endocrinology Metabolism and Hypertension, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No